CLINICAL TRIAL: NCT05226403
Title: Descriptive Study of Clinical and Pulmonary Ultrasound Signs of Acute Respiratory Infections Associated With COVID-19 in Primary Care
Brief Title: COVID-19 : Pulmonary Ultrasound in Primary Care
Acronym: ECHOVID-MG
Status: Completed | Type: Observational
Sponsor: Geprovas (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A01225-34
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Pulmonary Infection; Ultrasound Therapy; Complications; Respiratory Infection
Keywords: COVID19
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 infection are characterized by fever and signs of acute respiratory infection. A worsening of respiratory symptoms that can lead to respiratory failure. The decompensation can then be brutal and require rapid recourse to respiratory assistance. The contribution of clinical examination (auscultation and monitoring of oxygen saturation in particular) remains unsatisfactory in predicting an unfavorable course. The interest of pulmonary ultrasound is known in the management of pulmonary infections. However, estimating the severity of lung damage at an early stage could be of great help in monitoring and caring for patients. Ultrasound could meet this need in general practice, the chest scanner is often unavailable in these situations.

Ultrasound signs are associated with severe forms. The contribution of pulmonary ultrasound seems particularly interesting in the context of the reassessment of patients during the worsening phase of symptoms (D5-D10).

Estimate the prevalence of ultrasound signs in patients with an acute respiratory infection suspected or confirmed to be COVID-19, at the time of the worsening phase (between D5 and D10 of the onset of symptoms).

The prevalence of ultrasound lung lesions under COVID-19 may be essential to consider the development of the ultrasound tool in primary care. Indeed, if the contribution of ultrasound is now recognized in intensive care or emergency, its place in general medicine still raises questions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age with :

   * a clinical symptomatology suggesting an acute respiratory infection linked to COVID-19 defined by the following two categories of symptoms:

     * Sudden fever (or a feeling of fever)
     * Respiratory signs (cough, dyspnea, chest tightness) Or
   * an acute respiratory infection confirmed to COVID-19 by the result of RT-PCR screening tests.
2. And presenting, at the time of inclusion between the 5th and 10th day of infection, one of the respiratory signs of severity felt:

   * Dyspnea, shortness of breath or difficulty in breathing
   * Chest pain or tightness

Exclusion Criteria:

1. The presence of a severe form during the initial consultation. A severe form is defined by the presence of the following signs:

   * Polypnea> 22 / min
   * systolic BP <90 mmHg
   * Sp02 <90%
   * Altered consciousness, confusion, drowsiness
   * Dehydration
   * Alteration of the general condition in the elderly
2. The presence of acute respiratory signs clearly having a cause other than a COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with acute respiratory infection linked to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Ultrasound Signs | Between day 5 and day 10 of infection
  Frequency of the presence of at least one ultrasound sign in the subjects included

SECONDARY OUTCOMES:
Clinical Signs | Day 5 and Day 10
  Clinical signs positives in the cas of presence one of these elements: Hypoxia, Tachypnée, Pathological pulmonary auscultation.
Ultrasound signs | Between day 5 and day 10
  Ultrasound signs positives in the case of presence one of these elements: Disappearance of lines A, Appearance of three lines B, Appearance of pulmonary condensation.
Evolution and complication | Day 14 of infection
  Number of deaths and patients admitted to hospital for worsening of respiratory signs of infection

CONTACTS AND LOCATIONS:
Locations (1):
- GEPROVAS, Strasbourg, France